CLINICAL TRIAL: NCT02462889
Title: A Prospective, Single-Blind, Randomized Study to Evaluate Intravitreal Aflibercept Injection (IAI) Versus Sham as PROphylaxis Against CONversion to Neovascular Age-Related Macular Degeneration (AMD) in High-Risk Eyes
Brief Title: IAI Versus Sham as Prophylaxis Against Conversion to Neovascular AMD
Acronym: PRO-CON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jeffrey S Heier (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Jeffrey S Heier, Director, Vitreoretinal Service, Ophthalmic Consultants of Boston
Organization: Ophthalmic Consultants of Boston (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VGFTe-AMD-1507
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravitreal aflibercept injection (Experimental): Subjects will be randomized to receive intravitreal aflibercept injection every three months for 24 months.
  Interventions: Drug: Intravitreal aflibercept injection
- Placebo (Placebo Comparator): Subjects will be randomized to receive sham injection every three months for 24 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intravitreal aflibercept injection — Intravitreal aflibercept injection
  Other Names: Eylea
  Arms: Intravitreal aflibercept injection
Drug: Placebo — Sham injection
  Other Names: Sham injection
  Arms: Placebo

SUMMARY:
This is a prospective, single-blind, randomized study to evaluate intravitreal aflibercept injection (IAI) versus sham as prophylaxis against conversion to neovascular age-related macular degeneration (AMD) in "high-risk" subjects.

DETAILED DESCRIPTION:
128 subjects will be enrolled in the trial and randomized in a 1:1 ratio to receive either IAI every three months for 24 months or sham injections. Enrollment will be stratified in order to ensure a balance between the two treatment groups for subjects who were diagnosed with exudative AMD within the past two years versus those diagnosed more than two years prior to Baseline.

Study assessments will be conducted at required visits every three months and include manifest refraction and ETDRS visual acuity testing, slit lamp exam and dilated fundus exam, spectral-domain optical coherence tomography (SD-OCT) using Avanti device, and OCT angiography using Avanti AngioVueTM, and fluorescein angiography. Fundus photography will also be performed at Baseline, Month 12 and Month 24 visits.

In the event of conversion to neovascular AMD in the study eye at any point during the study, the Investigator will treat the subject with IAI at a frequency per his/her discretion.

ELIGIBILITY:
Inclusion Criteria:

* Study eye must have a diagnosis of non-exudative age-related degeneration characterized by the presence of many intermediate sized drusen, 1 or more large drusen, and/or hyperpigmentary changes. Fellow (non-study) eye must have CNV lesion (i.e., leakage on fluorescein angiography and/or subretinal, intraretinal, or sub-RPE fluid on OCT) secondary to age-related macular degeneration OR history of CNV lesion secondary to age-related macular degeneration, as confirmed by current or past treatment or current or past diagnostic imaging.
* Subject must be willing and able to comply with clinic visits and study-related procedures.
* Subject must provide signed informed consent.
* Subject must be able to understand and complete study-related questionnaires. In order to participate in the home monitoring sub-study, subjects must have an approved wireless device (i.e. iPhone, iPad, or iPod running iOS 6.0 or later) or be willing to use a loaned device and have access to a wireless Internet connection for the duration of the study.

Exclusion Criteria:

* Evidence of neovascular AMD in the study eye at time of enrollment or anytime in the past. The reading center must confirm that there is no evidence of neovascular AMD in the study eye prior to enrollment.
* Serous PED of any size in the study eye, as determined by the reading center.
* Previous treatment with verteporfin PDT, anti-VEGF therapy, laser, external beam radiation or other AMD therapy in the study eye.
* History of macular hole in study eye.
* History of vitrectomy in study eye.
* Lens extraction or implantation within the last 3 months.
* Capsulotomy within the last 1 month.
* Lens or other media opacity that would preclude good fundus photography or angiography within the next 2 years.
* Macular edema or signs of diabetic retinopathy more severe than 10 red dots (microaneurysms or blot hemorrhages).
* Retinal changes related to high myopia and/or myopic correction greater than 8.00 diopters spherical equivalent.
* Any progressive ocular disease that would affect visual acuity within the next 2 years.
* Previous participation in any studies of investigational drugs likely to have ocular effects within 30 days preceding the initial study treatment.
* Concurrent use of systemic anti-VEGF agents.
* Active or recent (within 4 weeks) intraocular inflammation (grade trace or above) in the study eye.
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye.
* For subjects who have undergone prior refractive or cataract surgery in the study eye, the preoperative refractive error in the study eye cannot exceed 8 diopters of myopia.
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure greater than 25 mmHg) despite treatment with anti-glaucoma medication).
* Subjects who are unable to be photographed to document CNV due to known allergy to fluorescein dye, lack of venous access or cataract obscuring the CNV.
* Subjects with other ocular diseases that can compromise the visual acuity of the study eye such as amblyopia and anterior ischemic optic neuropathy.
* Current treatment for active systemic infection.
* Evidence of significant uncontrolled concomitant diseases such as cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine, or gastrointestinal disorders.
* History of recurrent significant infections or bacterial infections.
* Inability to comply with study or follow-up procedures.
* Pregnancy (positive pregnancy test) or lactation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Heier, MD, Principal Investigator — Ophthalmic Consultants of Boston
Locations (4):
- United States (4):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - NJ Retina, Edison, New Jersey
  - Retina Consultants of Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heier JS, Brown DM, Shah SP, Saroj N, Dang S, Waheed NK, Wykoff CC, Prenner JL, Boyer DS. Intravitreal Aflibercept Injection vs Sham as Prophylaxis Against Conversion to Exudative Age-Related Macular Degeneration in High-risk Eyes: A Randomized Clinical Trial. JAMA Ophthalmol. 2021 May 1;139(5):542-547. doi: 10.1001/jamaophthalmol.2021.0221. PMID 33734306

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 128 patients enrolled, 127 (63 in the IAI group and 64 in the sham group) were included in the analysis. This is because shortly after enrollment of the excluded patient, it was determined that they should not have been enrolled due to not meeting eligibility criteria at screening.
Period: Overall Study
Arm/Group | Intravitreal aflibercept injection | Placebo
Started | 63 | 64
Completed | 60 | 53
Not Completed | 3 | 11
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Death | 1 | 5

BASELINE CHARACTERISTICS:
Population: 1 patient in Intravitreal aflibercept injection group had exudative disease in the study eye at Baseline, which was exclusionary.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravitreal Aflibercept Injection | Placebo | Total
Number analyzed (Participants) | 63 | 64 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.1 (7.4) | 76.9 (8.8) | 76.5 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 32 | 59
  Male | 36 | 32 | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Duration of Fellow Eye nvAMD < 2 Years [Count of Participants; unit: Participants] | 30 | 31 | 61
Non-exudative Macular NV [Count of Participants; unit: Participants] | 4 | 6 | 10
Mean BCVA [Mean (Standard Deviation); unit: letters read on ETDRS eye chart] — BCVA is best-corrected visual acuity. It is evaluated by counting the number of letters correctly read by the patient on an ETDRS eye chart. A higher value indicates that the patient read more letter correctly which indicates a better outcome.
  letters read on ETDRS eye chart | 78.7 (8.8) | 77.3 (10.1) | 78.0 (9.45)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Converting to Exudative AMD at 24 Months.
Description: Percentage of subjects converting to exudative AMD at 24 months as confirmed by independent masked reading center.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intravitreal aflibercept injection | Placebo
Number analyzed (Participants) | 63 | 64
Participants | 6 | 7

2. Secondary Outcome: Percentage of Patients Converted to Exudative AMD Who Had Exudative AMD in Fellow Eye ≤ 2 Years at Baseline.
Description: Percentage of patients converted to exudative AMD in study eye who had exudative AMD in fellow eye ≤ 2 years at Baseline.
Time Frame: up to Month 24
Population: Patients with a history of exudative AMD in their fellow eye no longer than 2 years at Baseline by treatment group.
Measure: Count of Participants; unit: Participants
Groups:
- Intravitreal Aflibercept Injection: Patients with a history of exudative AMD in their fellow eye of no longer than 2 years.
- Placebo: Patients with a history of exudative AMD in their fellow eye no longer than 2 years.
Arm/Group | Intravitreal Aflibercept Injection | Placebo
Number analyzed (Participants) | 30 | 31
Participants | 4 | 5

3. Secondary Outcome: Percentage of Patient Converted to Exudative AMD Based on Presence of Nonexudative CNV.
Description: Percentage of patients converted to exudative AMD compared to all patients with presence of nonexudative CNV in the study eye at Month 24, as confirmed by independent reading center evaluation of OCT angiography images.
Time Frame: up to Month 24
Population: Number of subjects with nonexudative CNV present at Month 24 based on OCT angiography.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravitreal aflibercept injection | Placebo
Number analyzed (Participants) | 11 | 13
Participants | 3 | 4

4. Secondary Outcome: Mean Change in Best-corrected Visual Acuity at 24 Months Compared to Baseline
Description: Mean change in best-corrected visual acuity (BCVA) at 24 months compared to baseline according to ETDRS protocol. BCVA is evaluated by counting the number of letters correctly read by the patient on an ETDRS eye chart. A higher value indicates that the patient read more letter correctly which indicates a better outcome.
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: number of letters read on eye chart
Arm/Group | Intravitreal aflibercept injection | Placebo
Number analyzed (Participants) | 63 | 64
number of letters read on eye chart | 2.8 [0.70 to 6.64] | 0.2 [-4.39 to 2.52]

5. Secondary Outcome: Mean Change in Growth of Geographic Atrophy.
Description: Mean change in growth of geographic atrophy from baseline to Month 24.
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: millimeters squared
Arm/Group | Intravitreal aflibercept injection | Placebo
Number analyzed (Participants) | 63 | 64
millimeters squared | 0.34 [-0.07 to 0.36] | 0.43 [0.11 to 0.96]

ADVERSE EVENTS:
Time Frame: 2 years
Description: A SAE is any untoward medical occurrence that at any dose:
  * Results in death.
  * Is life threatening.
  * Requires in-patient hospitalization or prolongation of existing hospitalization.
  * Results in persistent or significant disability/incapacity.
  * Is an important medical event. Events with severity score of Severe on 3-point scale of mild, moderate, or severe are reported.
Arm/Group | Intravitreal aflibercept injection | Placebo
All-Cause Mortality (participants affected / at risk) | 1/63 | 5/64
Serious Adverse Events (participants affected / at risk) | 14/63 | 27/64
Other Adverse Events (participants affected / at risk) | 9/63 | 8/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravitreal aflibercept injection (N=63) | Placebo (N=64)
Acute renal failure (Renal and urinary disorders) | 0 | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 | 1 (1)
Bleeding duodenum erosion (Gastrointestinal disorders) | 0 | 1 (1)
Blood loss from fall requiring transfusion (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Carcinoma in situ of the vulva (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Congestive heart failure (Cardiac disorders) | 0 | 1 (1)
CVA (Vascular disorders) | 1 (1) | 3 (3)
Elective cardioversion (Cardiac disorders) | 0 | 1 (1)
Fractured femur (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Gastric antral ulcer bleeding (Gastrointestinal disorders) | 0 | 1 (1)
Hip replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (3)
Infection right elbow (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Internal bleeding (Gastrointestinal disorders) | 0 | 2 (2)
Intestinal adhesions (Gastrointestinal disorders) | 0 | 1 (2)
Irregular heartbeat (Cardiac disorders) | 1 (1) | 0
Lung cancer (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Metastatic prostate cancer (Reproductive system and breast disorders) | 1 (1) | 0
Pleural effusion & dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (5)
Pulmonary edema due to failed heart valve (Cardiac disorders) | 1 (1) | 0
Right hip arthroplasty (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
RSV infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Subarachnoid hemorrhage (Nervous system disorders) | 0 | 1 (1)
Subdural hematoma (Nervous system disorders) | 0 | 1 (1)
Syncope due to fast VT or VF (Cardiac disorders) | 0 | 1 (1)
Tracheal cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravitreal aflibercept injection (N=63) | Placebo (N=64)
Abdominal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Decreased visual acuity x 6 lines (Eye disorders) | 1 (1) | 0
Elevated LFTs (Hepatobiliary disorders) | 1 (1) | 0
Hematochezia (Gastrointestinal disorders) | 0 | 1
Left cavernous sinus lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Leg pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Lump in right breast (Reproductive system and breast disorders) | 1 (1) | 0
Meniscus tear, left (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Nosebleed (Vascular disorders) | 0 | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Syncopal episode due to hypotension (Cardiac disorders) | 0 | 1 (1)
Thyroid nodule, benign (Endocrine disorders) | 0 | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0
Vulva intraepithelial neoplasia (VIN 3) (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Worsening of cataract (Eye disorders) | 0 | 1 (1)

LIMITATIONS AND CAVEATS:
No limitations. Trial was completed as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT02462889/Prot_SAP_000.pdf